CLINICAL TRIAL: NCT03473730
Title: A Pilot Study of Daratumumab (CD38 Antagonist) in Patients with Metastatic Renal Cell Carcinoma or Muscle Invasive Bladder Cancer
Brief Title: Daratumumab in Treating Patients with Muscle Invasive Bladder Cancer or Metastatic Kidney Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen Research & Development, LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0688; NCI-2018-00800 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0688 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Bladder Urothelial Carcinoma; Clear Cell Renal Cell Carcinoma; Malignant Urinary System Neoplasm; Metastatic Kidney Carcinoma; Stage IV Renal Cell Cancer AJCC V8
MeSH Terms: conditions — Carcinoma, Renal Cell; Urologic Neoplasms | interventions — Biopsy; daratumumab; Metastasectomy; Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 Renal (daratumumab, biopsy, surgery) (Experimental): Patients receive daratumumab IV over 8 hours for the first dose and then over 4 hours for all doses thereafter during weeks 1-8. Treatment repeats every week for up to 8 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo biopsy, nephrectomy, or metastasectomy during weeks 10-12. Patients may then restart treatment with daratumumab beginning 2 weeks after biopsy or 4-6 weeks after nephrectomy or metastasectomy. Cycles repeat every 2 weeks for 4 months and then monthly for 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Biological: Daratumumab; Other: Laboratory Biomarker Analysis; Procedure: Metastasectomy; Procedure: Nephrectomy
- Cohort 2 Bladder (daratumumab) (Experimental): Patients receive daratumumab IV over 8 hours for the first dose and then over 4 hours for all doses thereafter beginning at week 1. Cycles repeat every week for up to 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx
  Arms: Cohort 1 Renal (daratumumab, biopsy, surgery)
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Metastasectomy — Undergo metastasectomy
  Arms: Cohort 1 Renal (daratumumab, biopsy, surgery)
Procedure: Nephrectomy — Undergo nephrectomy
  Arms: Cohort 1 Renal (daratumumab, biopsy, surgery)

SUMMARY:
Objectives:

Primary:

Safety and tolerability of therapy with daratumumab in a cohort of patients with metastatic renal cell carcinoma and a cohort of patients with muscle invasive bladder cancer.

Secondary:

1A. To assess the proportion of patients who achieve pathological CR with daratumumab in patients with muscle invasive bladder cancer.

1B. To assess the objective response rate (ORR) to daratumumab in patients with metastatic renal cell carcinoma.

2. To assess the progression free survival for patients with metastatic renal cell carcinoma receiving Daratumumab.

DETAILED DESCRIPTION:
Detailed Description:

Bladder Cancer Cohort:

Study Drug Administration:

If you are eligible and agree to take part in this study, you will receive daratumumab by vein 1 time each week for 4 weeks before your cystectomy. During Week 1, your dose of daratumumab will be given over 8 hours. After that, each dose will be given over about 4 hours.

In this study, the following will be done to lower the chance of a daratumumab infusion related reaction:

You will get drugs, including steroids, acetaminophen, and/or antihistamine before the infusion. If you are considered high risk, you may also get drugs, including inhaled steroids, after the infusion.

The infusion may be slowed down or stopped if you have a reaction. You may stay overnight in the hospital after the infusion so the study staff can check your health.

You may ask the study staff for more information about the types of medications you will receive to lower your chance of an infusion-related reaction, including how they are administered and their risks.

Length of Study:

You may receive up to 4 doses of daratumumab before your surgery. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visit (described below).

Study Visits:

During Weeks 1-4:

You will have a physical exam. Blood (about 2 tablespoons) will be drawn for routine and blood type testing. Daratumumab will interfere with blood type testing which is needed before blood transfusions can be given. For this reason, a test to find out your blood type will be performed before you receive daratumumab. You should carry the blood type card with you while you are on this study.

During Weeks 6-8 (the week of your surgery):

You will have a physical exam. Blood (about 2 tablespoons) will be drawn for routine tests and part of this sample will also be used for blood type testing.

You will have surgery to remove your bladder. You will sign a separate consent form explaining the procedure and its risks in more detail.

End-of-Study Visit:

During Weeks 12-14, blood (about 2 tablespoons) will be drawn for routine tests.

Follow-Up Visit:

During Week 18, blood (about 2 tablespoons) will be drawn for routine tests and you will be asked about any side effects you are having.

Renal Cancer Cohort:

Study Drug Administration:

If you are eligible and agree to take part in this study, you will receive daratumumab by vein 1 time each week for 8 weeks before your nephrectomy, metastasectomy, or biopsy. During Week 1, your dose of daratumumab will be given over 8 hours. After that, each dose will be given over about 4 hours.

In this study, the following will be done to lower the chance of a daratumumab infusion related reaction:

You will get drugs, including steroids, acetaminophen, and/or antihistamine before the infusion. If you are considered high risk, you may also get drugs, including inhaled steroids, after the infusion.

The infusion may be slowed down or stopped if you have a reaction. You may stay overnight in the hospital after the infusion so the study staff can check your health.

You may ask the study staff for more information about the types of medications you will receive to lower your chance of an infusion-related reaction, including how they are administered and their risks.

Length of Study:

You may receive up to 8 doses of daratumumab prior to your surgery or biopsy. You may receive additional doses of daratumumab after the surgery/biopsy for up to one year after your first dose. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visit (described below).

Study Visits:

During Weeks 1-8:

You will have a physical exam each week before you receive daratumumab. Blood (about 2 tablespoons) will be drawn for routine and blood type testing. Daratumumab treatment will interfere with blood type testing which is needed before blood transfusions can be given. For this reason, a test to find out your blood type will be performed before you receive daratumumab. You should carry the blood type card with you while you are on this study.

During Weeks 10-12 (the week of your surgery/tissue collection):

You will have a physical exam. Blood (about 2 tablespoons) will be drawn for routine tests, part of this sample will also be used for blood type testing.

You will have surgery to remove your kidney, a kidney cancer lesion, or repeat biopsy. You will sign a separate consent form explaining the procedure and its risks in more detail.

During Weeks 14-30:

You will have a physical exam and return every 2 weeks to receive daratumumab. Blood (about 2 tablespoons) will be drawn for routine and blood type testing.

During Weeks 30-52:

You will have a physical exam and return every month to receive daratumumab. Blood (about 2 tablespoons) will be drawn for routine and blood type testing.

End-of-Study Visit:

During Week 52, blood (about 2 tablespoons) will be drawn for routine tests.

Follow-Up Visit:

During Week 65, blood (about 2 tablespoons) will be drawn for routine tests and you will be asked about any side effects you are having.

ELIGIBILITY:
Inclusion Criteria:

* RENAL & BLADDER COHORT: Consent to Monroe Dunaway (MD) Anderson laboratory protocol PA13-0291
* RENAL COHORT: Histological documentation of renal cell carcinoma with a clear cell component in the metastatic renal cell carcinoma cohort
* RENAL COHORT: Patients with an outside biopsy within 12 months is allowed for entry requirements; during the screening phase, patients without a tissue diagnosis may undergo a renal biopsy for histologic confirmation on PA13-0291
* RENAL COHORT: Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria in at least one site that is not the site for planned surgical resection or serial biopsy
* RENAL COHORT: If the kidney primary tumor is in place this is the preferred site of biopsy
* RENAL COHORT: Patients who have progression of disease or intolerance to a tyrosine kinase inhibitor (TKI) and to a PD-1 (like nivolumab) or PD-L1 (like atezolizumab) regimen; there is no limit to number of prior treatment regimens as long as the patient meets other eligibility criteria
* RENAL & BLADDER: Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s)
* RENAL & BLADDER: Female subjects of childbearing potential must not be pregnant at screening; females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy); however, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons
* RENAL & BLADDER: Eastern Cooperative Oncology Group (ECOG) performance status (PS) grade of =< 2
* RENAL COHORT: Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 from toxicities related to any prior treatments, unless adverse events (AEs) are clinically nonsignificant and/or stable on supportive therapy
* RENAL COHORT: Absolute neutrophil count (ANC) >= 1500/mm^3 without colony stimulating factor support (within 4 days before the first dose of daratumumab)
* RENAL COHORT: Platelets >= 100,000/mm^3 (within 4 days before the first dose of daratumumab)
* RENAL COHORT: Hemoglobin >= 9 g/dL (within 4 days before the first dose of daratumumab)
* RENAL COHORT: Bilirubin =< 1.5 x upper limit of normal (ULN); for subjects with known Gilbert's disease, bilirubin =< 3.0 mg/dL (within 4 days before the first dose of daratumumab)
* RENAL COHORT: Serum albumin >= 2.8 g/dl (within 4 days before the first dose of daratumumab)
* RENAL COHORT: Serum creatinine clearance (CrCl) >= 20 mL/min (within 4 days before the first dose of daratumumab); dialysis patients will be excluded; for creatinine clearance estimation, the Cockcroft and Gault equation should be used
* RENAL COHORT: Serum phosphorus >= lower limit of normal (LLN) (within 4 days before the first dose of daratumumab)
* RENAL COHORT: Calcium >= LLN (within 4 days before the first dose of daratumumab)
* RENAL COHORT: Magnesium >= LLN (within 4 days before the first dose of daratumumab)
* RENAL COHORT: Potassium >= LLN (within 4 days before the first dose of daratumumab)
* RENAL & BLADDER: Each subject must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures required for the study and is willing to participate in the study
* BLADDER: Histological documentation of urothelial cancer either on outside transurethral bladder biopsy or on initial transurethral bladder biopsy at MD Anderson under PA13-0291
* BLADDER: Patients may not have evidence of metastatic disease on baseline computed tomography (CT) or magnetic imaging resonance of the chest, abdomen, or pelvis
* BLADDER: Patients must be considered to be an operative candidate by the urology service at MD Anderson Cancer Center
* BLADDER: The patient must be systemic treatment naive, previous intra-vesicle therapy is allowed
* BLADDER: Subjects must be considered cisplatin ineligible as per treating physician due to renal dysfunction, hearing impairment, or co-morbidities; cisplatin ineligibility defined as: glomerular filtration rate (GFR) less than 60; congestive heart failure (CHF) New York Heart Association (NYHA) class III or higher; peripheral neuropathy grade 2 or higher; ECOG PS 2 or higher; impaired hearing
* BLADDER: ANC >= 1500/mm^3 without colony stimulating factor support (clinical laboratory values at screening)
* BLADDER: Platelets >= 100,000/mm^3 (clinical laboratory values at screening)
* BLADDER: Hemoglobin >= 9 g/dL (clinical laboratory values at screening)
* BLADDER: Bilirubin =< 1.5 x the ULN; for subjects with known Gilbert's disease, bilirubin =< 3.0 mg/dL (clinical laboratory values at screening)
* BLADDER: Serum albumin >= 2.8g/dl (clinical laboratory values at screening)
* BLADDER: Serum creatinine clearance (CrCl) >= 20 mL/min (clinical laboratory values at screening); dialysis patients will be excluded; for creatinine clearance estimation, the Cockcroft and Gault equation should be used
* BLADDER: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x ULN (clinical laboratory values at screening)
* BLADDER: Each subject must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures required for the study and is willing to participate in the study

Exclusion Criteria:

* RENAL & BLADDER: Currently enrolled in another interventional study
* RENAL COHORT: The subject has received any other type of investigational agent within 28 days before the first dose of study treatment
* RENAL COHORT: Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 2 weeks before the first dose of study treatment; eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of study treatment
* RENAL & BLADDER: Known evidence of an active infection requiring systemic therapy such as human immunodeficiency virus (HIV), active hepatitis, or fungal infection
* RENAL & BLADDER: History of clinically significant cardiovascular disease including, but not limited to:

  * Myocardial infarction or unstable angina =< 6 months prior to treatment initiation
  * Clinically significant cardiac arrhythmia
  * Deep vein thrombosis, pulmonary embolism, stroke =< 6 months prior to treatment initiation
  * Congestive heart failure (New York Heart Association class III-IV)
  * Pericarditis/clinically significant pericardial effusion
  * Myocarditis
  * Endocarditis
* RENAL & BLADDER: Other prior malignancy (exceptions: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) =< 2 years prior to enrollment
* RENAL & BLADDER: Any condition that in the opinion of the investigator, would preclude participation in this study
* RENAL & BLADDER: Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]); subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [antiHBc] and/or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels; those who are PCR positive will be excluded; EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR; seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 weeks after completion of study treatment (bladder cohort) or 6 weeks post-surgery (renal cohort)
  Adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will be recorded for all patients, recording name, grade, start and end dates, attribution to study drug, and whether the event was alleviated or controlled with relevant appropriate care similar to Phase I trials. Adverse events, serious adverse events (SAEs), and toxicities (TOX) will be summarized by grade and attribution in descriptive tables and figures by cohort.
Rate of surgical delay (Bladder cohort) | Up to 2 weeks after completion of study treatment
  To be defined as a delay greater than 4 weeks from planned intervention (week 10-12).
Incidence of surgical complications (Bladder cohort) | At 30 days post-surgery

SECONDARY OUTCOMES:
Pathologic response (Bladder cohort) | Up to 2 weeks after completion of study treatment
  Pathologic complete response (CR) (pCR) is defined as the absence of residual tumor in the radical cystectomy specimen and pelvic lymph node dissection (ie, ypT0N0). Patients who do not undergo surgery for any reason will be counted as not having a pCR. pCR rates and their 90% credible confidence intervals will be estimated using an uninformative beta distribution with a prior Beta (1,1).
Best objective response rate (ORR) (Renal cohort) | Up to 2 weeks after completion of study treatment
  ORR will be defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. Patients who have CR or partial response (PR) will be counted as having an objective response. ORR rates and their 90% credible confidence intervals will be estimated using an uninformative beta distribution with a prior Beta (1,1).
Progression-free survival (PFS) (Renal cohort) | From the start of study treatment up to 6 weeks post-surgery
  PFS will be defined as the time from first treatment to progression or death, regardless of cause, whichever comes first. Patients who are alive and free of progression at the time of data lock will be censored on the date they were last assessed for disease status (last follow-up). Patients who start a new therapy without progression will be censored on their last follow-up before starting the subsequent therapy. PFS will be estimated by Kaplan-Meier estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Campbell, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org